CLINICAL TRIAL: NCT03682666
Title: The Clinical Effect and Sonographic Findings of Kinesiotaping and Constraint Induced Movement Therapy in Upper Extremity Function and Spasticity in Patients With Subacute Stroke
Brief Title: Kinesiotaping and Constraint Induced Movement Therapy in Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMRPG8H0701
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: stroke; Kinesiotaping; constraint induced movement therapy; sonography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KT group (Active Comparator): the patients will perform Kinesiotaping for 5 days per week for 3 weeks
  Interventions: Device: Kinesiotaping
- mCIMT group (Sham Comparator): the unaffected limb will be constraint for 2 hours a day, 5 days a week for three weeks.
  And they will receive sham taping on the affected limb.
  Interventions: Behavioral: modified Constraint Induced Movement Training; Device: Sham taping
- KT+mCIMT group (Experimental): the patients will perform Kinesiology taping for 5 days per week for 3 weeks, and while being taped, the modified Constraint Induced Movement Training would be also executed.
  Interventions: Device: Kinesiotaping; Behavioral: modified Constraint Induced Movement Training

INTERVENTIONS:
Device: Kinesiotaping — Kinesio tape would be applied over the extensor muscles of the affected hand for facilitating the extension of hand. We will apply the tape from the upper 1/3 length of dorsal side of the forearm and split the tape into five equal bars to the distal interphalangeal joint of each finger along the finger bones. This intervention would be executed for five days per week for three weeks.
  Arms: KT group; KT+mCIMT group
Behavioral: modified Constraint Induced Movement Training — A 2-hour time period would be arranged to constraint patient's unaffected hand by using a bandage by a therapist. During this two hours, patients would not be allowed to use this unaffected to do any activity, so that they will need to use the affected hand. The caregivers would also be educated to provide less help if it is not necessary. This intervention would be executed two hours a day for five days per week, for three weeks.
  Arms: KT+mCIMT group; mCIMT group
Device: Sham taping — A short piece of kinesio tape would be cut into half and applied over the lateral side of the forearm from the lateral epicondyle till the half of the forearm. The tape would not cover the both the flexor and extensor muscle bellies.
  Arms: mCIMT group

SUMMARY:
In stroke patients, the most common neurological deficits were motor impairment, loss of somatosensation, abnormal muscle tone, and impaired fractionated movement at affected limbs. Therefore, the investigators try to facilitate upper extremity function and normalize the muscle tone to enlarge their capacity to perform daily activities and to improve life quality by modified constraint-induced movement therapy (mCIMT) and Kinesiotaping (KT).

The investigators will collect 90 subacute stroke patients with hemiplegia in this study. These 90 patients will be randomly divided into 3 groups. In KT group (n=30), the patients will perform Kinesiology taping for 5 days per week for 3 weeks. In mCIMT group (n=30), the patient will receive constraint the unaffected limb for 2 hours a day, 5 days a week for three weeks. In KT+mCIMT group, the KT and mCIMT interventions would be performed for 5 days a week in three weeks. All the patients in KT, CIMT and KT+mCIMT groups will receive 20-minute hand function training twice daily for 5 days per week for 3 weeks. Before intervention, immediately and 3 week later after intervention, all patients will receive the physical examinations including motor recovery stage (Brunnstrom stage), spasticity (modified Ashworth scale and Tardieu scale), and sensation. Fugl-Meyer assessment for upper extremity (FMA-UE), box and block test, Simple Test for Evaluating Hand Function (STEF), and Wolf Motor Function Test for hand function, ADL and quality of life assessment and musculoskeletal sonography for affected forearms will be also evaluated in this study.

The aims of this study are:

1. To investigate the effect of Kinesiotaping and modified CIMT in improving upper extremity function and spasticity for subacute stroke patients with hemiplegia.
2. To explore the role of sonoelastography and shear wave velocity in poststroke spasticity assessment.

ELIGIBILITY:
Inclusion Criteria:

* The patients have a stroke with hemiplegia (duration is 3~12 months after stroke).
* Patients who are able to perform hand grasp.
* Patients who could slightly do fingers extension and minimal wrist extension. (ability of extension at least 10 degrees at the metacarpophalangeal and interphalangeal joints and 20 degrees at the wrist.)

Exclusion Criteria:

* age is younger than 18 years or older than 80 years
* previous history of upper extremity tendon or neuromuscular injury
* any other systemic neuromuscular disease
* cognition or language impairment leading to communication difficulty
* allergy history when application of KT materials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
the change from baseline to time of Fugl-Meyer assessment | 3rd week, and 6th week
  a therapist will evaluate Fugl-Meyer assessment for upper extremity (FMA-UE) for each participant. In this assessment, participants would need to execute a series of movements, which involved proximal and distal part of upper limb. The higher the grade, the better the performance.
the change from baseline to time of Musculoskeletal sonography | 3rd week, and 6th week
  an experienced physiatrist will evaluate the findings on sonography, sonoelastography, and shear wave velocity (SWV). The participants will sit upright and put their upper extremities on the bed with elbow flexion in 90 degrees and the forearm full supination. The measured levels for evaluating FCR, FCU, and FDS muscles will be recorded at first time and use the same level at follow up for each patient. The SWV will be done in the longitudinal/transverse planes and be performed at the maximal cross-section area of the muscles and repeatedly measured for 7 times for each muscle. The sonoelastography will be applied in the longitudinal plane of the detected muscles at the same level of the SWV.
the change from baseline to time of MAS scale | 3rd week, and 6th week
  a therapist will measure spasticity of affected upper extremity at elbow and wrist joints (modified Ashworth scale). In this scale, muscle tone would be assessed by quick stretch of muscle belly. The scoring criteria are as follows. 0, no increase in muscle tone; 1, Slight increase in muscle tone; 2, More marked increase in muscle tone through most of the ROM; 3, considerable increase in muscle tone; 4, affected part(s) rigid in flexion or extension.

SECONDARY OUTCOMES:
the change from baseline to time of Brunnstrom stage | 3rd week, and 6th week
  a therapist will measure motor recovery stage (Brunnstrom stage)
the change from baseline to time of modified Tardieu scale | 3rd week, and 6th week
  a therapist will measure spasticity of affected upper extremity at elbow and wrist joints (modified Tardieu scale).
the change from baseline to time of existence of sensation | 3rd week, and 6th week
  a therapist will measure the sensation, including light touch, pinprick touch, proprioception.
the change from baseline to time of quality of life by Stroke Impact Scale | 3rd week, and 6th week
  Stroke Impact Scale would be used to measure the independence of daily activities. It is a self-reported questionnaire. The contents involve various aspect of life. The high the grade, the more serious the life is affected.
the change from baseline to time of quality of life by Barthel Index | 3rd week, and 6th week
  Barthel Index would be used to measure the independence of daily activities. It is a form that contains different activities of daily living. The higher the outcome grades, the better the level of independence.
the change from baseline to time of functional performance by box and block test | 3rd week, and 6th week
  box and block test would be used to assess the grasping and release performance of the affected hand.
the change from baseline to time of functional performance by STEF | 3rd week, and 6th week
  Simple Test for Evaluating Hand Function (STEF) would be used to assess the hand function by executing various types of grasping.
the change from baseline to time of functional performance by Wolf Motor Function Test | 3rd week, and 6th week
  Wolf Motor Function Test would be used for measuring hand functions.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chi Huang, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No